CLINICAL TRIAL: NCT01877395
Title: Immunogenicity and Safety of the Purified Vero Rabies Vaccine - Serum Free in Comparison With the Rabies Human Diploid Cell Vaccine (Imovax® Rabies) Administered in a Simulated Rabies Post-exposure Regimen in Healthy Adults
Brief Title: Study of Purified Vero Rabies Vaccine and Rabies Human Diploid Cell Vaccine in a Simulated Rabies Post-exposure Regimen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VRV04; U1111-1117-7447 (Other: WHO)
Record Dates: First submitted 2013-06-10; First posted 2013-06-13 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-11

CONDITIONS: Rabies
Keywords: Rabies; Purified Vero Rabies Vaccine - Serum Free; Human Diploid Cell Vaccine; Imovax® Rabies
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Purified Vero Rabies Vaccine Group (Experimental): Participants will receive the Purified Vero Rabies Vaccine (VRVg)
  Interventions: Biological: Purified Vero Rabies Vaccine (VRVg)
- Imovax® Rabies Vaccine Group (Experimental): Participants will receive the Imovax® Rabies vaccine
  Interventions: Biological: Imovax® Rabies: inactivated rabies vaccine

INTERVENTIONS:
Biological: Purified Vero Rabies Vaccine (VRVg) — 0.5 mL, Intramuscular
  Arms: Purified Vero Rabies Vaccine Group
Biological: Imovax® Rabies: inactivated rabies vaccine — 1.0 mL, Intramuscular
  Other Names: Imovax® Rabies
  Arms: Imovax® Rabies Vaccine Group

SUMMARY:
The aim of the study is to document the safety and immunogenicity of Purified Vero Rabies Vaccine (VRVg) when given in a simulated post-exposure regimen, i.e. with co-administration of human rabies immunoglobulins (Imovax® Rabies).

Primary Objectives:

* To demonstrate that VRVg is non-inferior to Imovax® Rabies in terms of proportion of subjects achieving a rabies virus neutralizing antibody (RVNA) titer ≥ 0.5 international units (IU)/mL at Day 14.
* To demonstrate that the observed proportion of subjects achieving an RVNA titer ≥ 0.5 IU/mL at Day 14 is at least 99%, with a lower limit of the 95% confidence interval (CI) of at least 97%.

Secondary Objectives:

* To assess the clinical safety of each vaccine after each vaccine injection when administered in a simulated post-exposure schedule.
* To describe the geometric mean titer ratio (GMTR) between the 2 vaccine groups at Day 14.

DETAILED DESCRIPTION:
All participants will receive five vaccine injections, i.e. one at Day 0, at Day 3, at Day 7, at Day 14 and at Day 28, respectively, (Essen regimen). In addition, human rabies immunoglobulins (HRIG) will be concomitantly administered to all subjects on Day 0.

Safety will be assessed in all participants up to 28 days after vaccination, as applicable, in terms of occurrence of adverse events (AEs), and serious adverse events (SAEs) and adverse events of special interest (AESIs) up to 6 months post-vaccination 5.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to < 65 years on the day of inclusion
* Informed consent form has been signed and dated - Able to attend all scheduled visits and comply with all trial procedures.

Exclusion Criteria:

* Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination and until at least 4 weeks after the last vaccination)
* Participation at the time of study enrollment or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination or planned receipt of any vaccine during the course of the trial
* Previous vaccination against rabies (in pre- or post-exposure regimen) with either the trial vaccine or another vaccine
* Receipt of immunoglobulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Self-reported seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C
* At high risk of rabies infection during the trial
* Known systemic hypersensitivity to any of the components of either vaccine or HRIG, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances
* Self-reported thrombocytopenia, contraindicating intramuscular (IM) vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 100.4°F). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study
* History of Guillain-Barré Syndrome.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 342 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with rabies virus neutralizing antibody (RVNA) titer ≥ 0.5 IU/mL at Day 42 (14 days after the last vaccination of primary vaccination series). | Day 14 post-vaccination
  Rabies virus neutralizing antibody titer will be determined by the rapid fluorescent focus inhibition test (RFFIT)

SECONDARY OUTCOMES:
Number of Participants Reporting Solicited Injection Site Reactions, Solicited Systemic Reactions, Unsolicited Systemic Reactions, and Serious Adverse Events Occurring Throughout the Trial | Day 0 up to 6 months post-vaccination
  Solicited injection site reactions: pain, erythema, and swelling. Solicited systemic reactions: fever (temperature), headache, malaise, and myalgia.
Geometric mean titer ratio (GMTR) following vaccination with either Purified Vero Rabies Vaccine, Serum Free or Rabies Human Diploid Cell Vaccine in a Simulated Rabies Post exposure Regimen | Day 14 post-vaccination
  Rabies virus neutralizing antibody titer will be determined by the rapid fluorescent focus inhibition test (RFFIT)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (5):
- United States (5):
  - Pembroke Pines, Florida
  - South Miami, Florida
  - Boise, Idaho
  - Raleigh, North Carolina
  - West Jordan, Utah

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com